CLINICAL TRIAL: NCT06148571
Title: Left Bundle Branch Area Pacing in Heart Failure Patients With Ejection Fraction Below Normal
Status: Recruiting | Type: Observational
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Eue-Keun Choi, Professor, Seoul National University Hospital
Other Study IDs: LBBAP-HF
Record Dates: First submitted 2023-10-04; First posted 2023-11-28 (Actual); Last update posted 2025-05-18 (Actual); Status verified 2025-05

CONDITIONS: Left Ventricular Ejection Fraction Less Then or Equal to 50percent

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Prospective LBBAP-HF cohort: Patient who underwent attempted left bundle branch area pacing using Biotronik Selectra 3D sheath and stylet driven lead (Solia S60, Biotronik).
  Interventions: Device: left bundle branch area pacing
- Retrospective LBBAP-HF cohort: Patients who underwent attempted left bundle branch area pacing using Biotronik Selectra 3D and Solia S60 lead prior to prospective enrollment.
  Interventions: Device: left bundle branch area pacing

INTERVENTIONS:
Device: left bundle branch area pacing — left bundle branch area pacing locates ventricular lead into the interventricular septum to capture left bundle branch areas.

SUMMARY:
While cardiac resynchronization therapy remains the mainstay for advanced HF, it is not always feasible due to unfavorable anatomy of coronary sinus or pacing characteristics. In such cases, left bundle branch area pacing itself or left bundle optimized cardiac resynchronization therapy could be a rescue therapy for failed or unsuccessful biventricular cardiac resynchronization therapy. However, the efficacy and safety of left bundle branch area pacing (or left bundle optimized cardiac resynchronization therapy) as rescue therapy for biventricular cardiac resynchronization therapy is largely hypothetic and lack concrete evidence still.

Therefore, there is an unmet need for the registry purposed for left bundle branch area pacing among heart failure with mid-range (or mildly reduced) ejection fraction and heart failure with reduced ejection fraction patients to investigate its efficacy and safety.

This study aims to investigate the efficacy and safety of left bundle branch area pacing in heart failure patients with ejection fraction below normal using Selectra catheters.

ELIGIBILITY:
Inclusion Criteria:

* Patients previously diagnosed with heart failure with mid-range(or mildly reduced) ejection fraction and heart failure with reduced ejection fraction, which was documented by an appropriate echocardiographic study (Left ventricle ejection fraction <50%), and
* Patients with indications of cardiac pacing or cardiac resynchronization therapy

Exclusion Criteria:

* Patients aged less than 19 years.
* Pregnant.
* Patients with an expected life expectancy of less than 1 year.
* Patients with a mechanical valve for the tricuspid valve.
* Patients who need atrial pacing only.
* Patients who are not capable of receiving a transvenous pacemaker for any reason.

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who have EF below normal and require permanent cardiac pacing or CRT.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2023-10-10 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
The acute success rate of left bundle branch area pacing | The day of the procedure
  The acute success of left bundle branch area pacing was defined as below:
  Meet ≥2 criteria as follows evaluated at the end of the procedure.
  * Right bundle branch block configuration observed during unipolar tip pacing
  * Left bundle branch potential (Left bundle branch-Ventricular interval of 15 to 35ms)
  * Transition from nonselective Left bundle branch capture to selective Left bundle branch capture
  * Transition from nonselective Left bundle branch capture to left septal capture at near threshold outputs
  * Short and constant peak left ventricular activation time (stimulus to peak of the R wave in V5 or V6 [peak left ventricle activation time]) <75ms in non-Left bundle branch block and <85ms in Left bundle branch block
  Programmed (extra-stimulus testing) deep septal stimulation to differentiate left ventricular septal vs nonselective Left bundle branch capture
Acute complications related to the procedures | 7 days from the procedure
  * Death related to the procedure
  * Vascular complications (pocket hematoma, pseudoaneurysm, fistular, rupture)
  * Device-related infection
  * Cardiac perforation or tamponade
  * Septal perforation
  * Acute coronary syndrome
  * Pneumothorax, hemothorax
  * Thromboembolic events (stroke, pulmonary thromboembolism)
  * Lead dislodgment

SECONDARY OUTCOMES:
The incidence of acute procedure-related complication | 1 year
  The acute procedure-related complication was defined as the occurrence of the below-listed events within 7 days of the procedure.
  (Death related to the procedure, Pocket hematoma, Pseudoaneurysm, Fistular, Vascular rupture, Device-related infection, Cardiac perforation, Cardiac tamponade, Septal perforation, Acute coronary syndrome, Pneumothorax, Hemothorax, Stroke, Pulmonary thromboembolism, Lead dislodgement)
The incidence of repeat procedures | 1 year
  The incidence of repeat left bundle branch area pacing procedures
The incidence of pacemaker upgrade to cardiac resynchronization therapy including biventricular cardiac pacing | 1 year
  The incidence of pacemaker upgrade to cardiac resynchronization therapy including biventricular cardiac pacing
The incidence of heart failure hospitalization | 1 year
  The incidence of heart failure hospitalization
The incidence of cardiovascular death | 1 year
  The incidence of cardiovascular death
The incidence of All-cause death | 1 year
  The incidence of All-cause death
Left ventricular ejection fraction | 1 year
  Left ventricular ejection fraction (%)
Left ventricular end diastolic diameter | 1 year
  Left ventricular end diastolic diameter (mm)
Left ventricular end systolic diameter | 1 year
  Left ventricular end systolic diameter (mm)
left ventricular global strain | 1 year
  left ventricular global strain (%) if possible.
Capture threshold | 1 year
  Left bundle branch area pacing lead parameter: capture threshold (V)
Sensing | 1 year
  Left bundle branch area pacing lead parameter: sensing (mV)
Impedance | 1 year
  Left bundle branch area pacing lead parameter: impedance (Ohms)

CONTACTS AND LOCATIONS:
Overall Officials: Eue-Keun Choi, M.D. Ph.D., Principal Investigator — Seoul National University Hospital
Locations (1):
- Seoul National University Hospital, Seoul, Jongno-gu, South Korea

IPD SHARING:
Plan to Share IPD: Undecided